CLINICAL TRIAL: NCT05086367
Title: Effects of Breathing Exercises on Pain, Range of Motion and Neck Disability in Patients With Cervical Spondylosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-UOL-FAHS/770-1/2020
Record Dates: First submitted 2021-09-11; First posted 2021-10-20 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-09

CONDITIONS: Cervical Spondylosis
MeSH Terms: conditions — Spondylosis | interventions — Contraceptive Devices, Female

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine Physical Therapy (Active Comparator): This group received only routine physical therapy. This includes thermotherapy, trans-cutaneous electrical nerve stimulation, neck isometrics and stretching that includes 12 sessions (3 sessions per week)
  Interventions: Other: Routine Physical Therapy
- Breathing Exercises along with routine physical therapy (Experimental): This group received routine physical therapy along with breathing exercises. This includes thermotherapy, trans-cutaneous electrical nerve stimulation, neck isometrics and stretching that includes 12 sessions (3 sessions per week).
  Interventions: Other: Diaphragmatic and pursed lip breathing

INTERVENTIONS:
Other: Diaphragmatic and pursed lip breathing — Breathing exercises were performed. Two breathing techniques were applied to the participants. Diaphragmatic and pursed lip breathing were intervened along with routine physical therapy.
  Arms: Breathing Exercises along with routine physical therapy
Other: Routine Physical Therapy — Routine physical therapy exercises were performed in which neck isometrics and neck range of motion exercises were performed
  Arms: Routine Physical Therapy

SUMMARY:
A randomized controlled trial was conducted on 72 diagnosed patients with cervical spondylosis at University of Lahore Teaching hospital. The study was completed within 9 months after the approval of synopsis. Patients who fulfill the inclusion criteria were identified by individual physiotherapist and were enrolled for particular study. Informed written consent was be taken by the patients and were randomly allocated into two groups. The total numbers of sessions were 12 (3 sessions per week). The study was single blinded. The assessor was unaware of the treatment given to both groups.

Control group received only routine physical therapy. This includes thermotherapy, trans-cutaneous electrical nerve stimulation, neck isometrics and stretching that includes 12 sessions and three times per week.

Experimental group received routine physical therapy along with breathing exercises. This includes thermotherapy, trans-cutaneous electrical nerve stimulation, neck isometrics and stretching that includes 12 sessions and three times per week.

Baseline data was collected before first treatment then after 4th, 8th and 12th session.

The outcome measures were neck pain, ROM, neck disability and quality of life and were analyzed by using SPSS 26 and then results and conclusion were drawn.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed patients with cervical spondylosis
* Both male and female
* Age from 40-60 years

Exclusion Criteria:

* Any deformity of spine
* Any surgery of spine
* Tumor
* Trauma & Fracture
* Cervical radiculopathy
* Respiratory diseases

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2020-11-13 (Actual); Primary Completion 2021-08-07 (Actual); Study Completion 2021-09-07 (Actual)

PRIMARY OUTCOMES:
Change in Visual Analogue Scale score | Change from pre-intervention to 4 weeks
  Visual analogue scale was used to assess neck pain. Score ranges from 0-10. 0 shows least pain and 10 shows worst pain
Change in Universal Goniometer readings | Change from pre-intervention to 4 weeks
  Universal Goniometer was used to assess cervical range of motion.
Change in Neck Disability Index score | Change from pre-intervention to 4 weeks
  Neck Disability Index was used to assess neck disability. Score ranges from 0-50. 0 shows minimum disability and 50 shows maximum disability.

SECONDARY OUTCOMES:
Change in SF-36 Questionnaire score | Change from pre-intervention to 4 weeks
  SF-36 Questionnaire was used to assess quality of life. Scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Lahore Teaching Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No